CLINICAL TRIAL: NCT01984203
Title: Progressive Heavy Strength Training Compared to General Low-load Exercises in Patients With Rotator Cuff Tendinopathy: a Randomized Controlled Trial
Brief Title: Rotator Cuff Tendinopathy Exercise Trial
Acronym: RoCTEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other); Sygehus Lillebaelt (Other); Aalborg University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Kim Gordon Ingwersen, MSc, PhD.stud., University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RoCTExPRIMARY
Record Dates: First submitted 2013-10-31; First posted 2013-11-14 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Rotator Cuff Tendinitis
Keywords: Shoulder; Impingement; Rotator Cuff Syndrome; Subacromial Impingement Syndrome; Exercise; Physiotherapy
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Impingement Syndrome; Motor Activity | interventions — Exercise; Physical Therapy Modalities; Posture; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progressive Heavy Strength Exercises (Experimental): The Progressive Heavy Load Exercise group gradually increases the external load from 60%RM to 90%RM and correspondently decreases the number of performed repetitions pr. set for the two rotator cuff exercises. Furthermore 4 sets is performed.
  A progressive exercise program consisting of 6 active exercises. Two exercises for the rotator cuff: Full Can and Sidelying external rotation Two exercises for the scapulae stabilizing muscles: Low Row and Push-Up Plus Two glenohumeral/postural corrective exercises: Posterior GH stretch and Scapular Retraction.
  Interventions: Other: Progressive Heavy Strength Exercises
- Low Load Exercises (Active Comparator): Active exercises comparator continuously training with 60%RM through 12 weeks.
  An exercise program consisting of 6 active exercises. Two exercises for the rotator cuff: Full Can and Sidelying external rotation Two exercises for the scapulae stabilizing muscles: Low Row and Push-Up Plus Two glenohumeral/postural corrective exercises: Posterior GH stretch and Scapular Retraction.
  Interventions: Other: Low Load Exercises

INTERVENTIONS:
Other: Low Load Exercises — All rotator cuff and scapular exercises are performed with 3 sets of 20 repetitions 3 times per week for 12 weeks. The load is set at around 60% of 1 RM (20 reps).
  The glenohumeral/postural corrective exercises are performed with 3 sets of 5 repetitions (The position is held for 15 seconds per repetition).
  Other Names: Scapular stabilization; Rotator Cuff; Exercise; Physiotherapy; Posture; Progressive exercise; Strength training
  Arms: Low Load Exercises
Other: Progressive Heavy Strength Exercises — All scapular exercises are performed with 3 sets of 20 repetitions 3 times per week for 12 weeks. The load is set at around 60% of 1 RM (20 reps).
  The rotator cuff exercises are performed with 4 sets of gradually progressive loading and decreasing the repetitions performed in each set.
  Week 1: 15reps (70% 1RM) Week 2-3: 12 reps (75% 1RM) Week 4-5: 10 reps (80% 1RM) Week 6-8: 8 reps (85% 1RM) Week 9-12: 6 reps (90% 1RM)
  The glenohumeral/postural corrective exercises are performed with 3 sets of 5 repetitions (The position is held for 15 seconds per repetition).
  Other Names: Scapular stabilization; Rotator Cuff; Exercise; Physiotherapy; Posture; Progressive exercise; Strength training
  Arms: Progressive Heavy Strength Exercises

SUMMARY:
This study aims at determine if Progressive Heavy Load Exercises (PHLE) as treatment for patients diagnosed with Rotator Cuff Tendinopathy is superior to "Standard Low-Load Exercises" (LLE).

DETAILED DESCRIPTION:
The trial will be performed as a multicenter randomised controlled trail, including 110 patients diagnosed with Rotator Cuff Tendinopathy from four orthopaedic shoulder clinics in secondary sector in Denmark.

The PHLE intervention will consist of progressive strengthening exercises performed with heavy load dumbbells, targeting the rotator cuff in a 12 weeks home-exercise program with six control visits at a physiotherapy department at the hospitals.

The LLE exercise program consists of the same exercises as the PHLE, but performed with low load dumbbells.

"Disability of the Arm, Shoulder and Hand (DASH) questionnaire" is used as the primary outcome and is measured 12 weeks post baseline.

12 months post baseline a secondary follow-up will be performed primarily measuring the number of patients referred to an operation.

Patients will be randomised to either PHLE or LLE regime by blocks according to whether they have been referred to corticosteroid injection by their orthopaedic shoulder specialist.

*April 2015: (We originally expected to be able to include 260 patients in order to analyze our data according to the sub-groups of exercise group +/- Corticosteroid injection, but inclusion rate has been much lower then expected, and due to time restraints we only expect to include 110 patients)

Primary investigator and patients will be blinded towards group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years of age
* history of shoulder complaints lasting at least 3 months prior to enrolment
* Pain located in the proximal lateral aspect of the upper arm (C5 dermatome) aggravated by abduction
* Positive "Full Can test" AND/OR "Jobes test/Empty Can test" AND/OR "Resisted External Rotation test"
* Positive "Hawkins-Kennedy test AND/OR Neers test
* Ultra-sonographic verification of tendon swelling, hypo echoic areas, fibrillar disruption or neovascularization in the RC.

Exclusion Criteria:

* Resting pain more than 40 mm on a visual analogue scale (VAS);
* Bilateral shoulder pain
* Less than 90 degrees of active elevation of the arm;
* Full thickness RC rupture verified by ultra-sonography;
* Corticosteroid injection within the last 6 weeks;
* Radiologic verified fracture, calcification larger then 5 mm (vertical distance) in the RC tendon, glenohumeral arthrosis or malalignment in the shoulder complex;
* Prior surgery or dislocation of the affected shoulder;
* Clinically suspected labrum lesion, arthritis in the AC-joint, frozen shoulder or symptoms derived from the cervical spine;
* Sensory or motor deficit in neck or arm;
* Suspected competing diagnoses (e.g., Rheumatoid arthritis, Cancer, Neurological disorders, Fibromyalgia, Schizophrenia, Suicidal threatened, Borderline personality disorder, or Obsessive Compulsive Disorder);
* Pregnancy;
* Inability to fluently understand written and spoken Danish.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Disability of the Arm, Shoulder and Hand questionnaire at 12 weeks | Baseline and 12 weeks

SECONDARY OUTCOMES:
Change from baseline in Isometric Strength (MVC) | Baseline and 12 weeks
Change from baseline in Range of movement | Baseline and 12 weeks
Number of patients referred to or completed arthroscopic shoulder operation | 12 months
Change in Shoulder injury and Osteoarthritis Outcome Score - (SOOS) at 12 weeks | Baseline and 12 weeks
Hospital Anxiety and Depressions score - (HAD) | Baseline
Scapula Retraction test | Baseline
Scapula Assisted Test | Baseline
Change in Euro Qol 5D index (EQ 5D) at 12 weeks | Baseline and 12 weeks
Change in Disability of the Arm, Shoulder and Hand questionnaire at 52 weeks | Baseline and 52 weeks
Change in Shoulder injury and Osteoarthritis Outcome Score - (SOOS) at 52 weeks | Baseline and 52 weeks
Change in Euro Qol 5D index (EQ 5D) at 52 weeks | Baseline and 52 weeks

OTHER OUTCOMES:
Change in tendon quality measured on ultra-sonography at 12 weeks | Baseline and 12 weeks
Baseline demographic and Socioeconomic variables measured at 52 weeks | Baseline and 52 weeks
  Age, sex, duration of symptoms, symptom history, number of patients receiving corticosteroid injections, visits at the patients general practitioner related to their shoulder problem, visits at the secondary healthcare system related to their shoulder problem, sick leave

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Juul-Kristensen, Ass. Prof, Study Director — University of Southern Denmark
Locations (3):
- Denmark (3):
  - Odense University Hospital - Svendborg Hospital, Odense, Fyn
  - Aalborg University Hospital - Himmerland Hospital, Aalborg, Jutland
  - Hospital Lillebaelt - Vejle Hospital, Vejle, Jutland

REFERENCES:
- [Derived] Ingwersen KG, Jensen SL, Sorensen L, Jorgensen HR, Christensen R, Sogaard K, Juul-Kristensen B. Three Months of Progressive High-Load Versus Traditional Low-Load Strength Training Among Patients With Rotator Cuff Tendinopathy: Primary Results From the Double-Blind Randomized Controlled RoCTEx Trial. Orthop J Sports Med. 2017 Aug 28;5(8):2325967117723292. doi: 10.1177/2325967117723292. eCollection 2017 Aug. PMID 28875153
- [Derived] Ingwersen KG, Hjarbaek J, Eshoej H, Larsen CM, Vobbe J, Juul-Kristensen B. Ultrasound assessment for grading structural tendon changes in supraspinatus tendinopathy: an inter-rater reliability study. BMJ Open. 2016 May 24;6(5):e011746. doi: 10.1136/bmjopen-2016-011746. PMID 27221128
- [Derived] Ingwersen KG, Christensen R, Sorensen L, Jorgensen HR, Jensen SL, Rasmussen S, Sogaard K, Juul-Kristensen B. Progressive high-load strength training compared with general low-load exercises in patients with rotator cuff tendinopathy: study protocol for a randomised controlled trial. Trials. 2015 Jan 27;16:27. doi: 10.1186/s13063-014-0544-6. PMID 25622594
- See also: Protocol article — http://www.ncbi.nlm.nih.gov/pubmed/25622594